CLINICAL TRIAL: NCT04881994
Title: Investigation of the Pharmacokinetics, Safety, and Tolerability of Finerenone (BAY 94-8862) in Subjects With Hepatic Impairment (Classified as Child Pugh A or B) and in Age-, Weight-, and Gender-matched Healthy Subjects Following a Single Oral Dose in a Single-center, Non-randomized, Non-controlled, Non-blinded, Observational Study With Group Stratification
Brief Title: A Study to Learn How Finerenone (BAY94-8862) Moves Into, Through and Out of the Body, How it Affects the Body, and How Safe it is in Adult Participants With Different Degrees of Reduced Liver Function and in Healthy Participants With Similar Age, Weight and Gender Distribution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14510; 2013-005089-21 (EudraCT Number)
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Worsening Chronic Heart Failure; Diabetic Nephropathy
Keywords: Child Pugh A; Child Pugh B; Liver impairment
MeSH Terms: conditions — Diabetic Nephropathies | interventions — finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild hepatic impairment (Child Pugh A) (Experimental): Participants with mild hepatic impairment (Child Pugh A) received single oral dose of finerenone.
  Interventions: Drug: Finerenone (BAY94-8862)
- Moderate hepatic impairment (Child Pugh B) (Experimental): Participants with moderate hepatic impairment (Child Pugh B) received single oral dose of finerenone.
  Interventions: Drug: Finerenone (BAY94-8862)
- Healthy participants (Experimental): Healthy age-, weight-, and gender- matched participants received single oral dose of finerenone.
  Interventions: Drug: Finerenone (BAY94-8862)

INTERVENTIONS:
Drug: Finerenone (BAY94-8862) — Single oral dose of finerenone given as 5 mg immediate release (IR) tablet.

SUMMARY:
Researchers are looking for a better way to treat people who have worsening of chronic heart failure, a long-term condition where the heart does not pump blood as well as it should, as well as to treat patients who have diabetic nephropathy, a long-term, progressive decrease in the kidneys' ability to work properly in patients with diabetes mellitus.

In this study researchers wanted to learn more about a new substance called finerenone (BAY94-8862). Finerenone is a substance that blocks the activation of a protein in the body called mineralocorticoid receptor (MR). An increased activation of MR is involved in the development of hypertension, organ damage and worsening of heart failure.

The researchers studied how finerenone moves into, through and out of the body. The researchers also looked at how safe finerenone is and how it affects the body. The main purpose of this study was to help researchers develop recommendations for the amount of the substance (the dosing) to be given to patients with reduced liver function.

ELIGIBILITY:
Inclusion Criteria:

All participants

* The informed consent must be signed before any study specific tests or procedures are done;
* Male and female white participants;
* Women of childbearing potential can only be included in the study if a pregnancy test is negative. Women of childbearing potential must agree to use adequate contraception when sexually active. 'Adequate contraception' is defined as any combination of at least 2 effective methods of birth control, of which at least one is a physical barrier (e.g. condoms with hormonal contraception or implants or combined oral contraceptives, certain intrauterine devices). This applies from signing the informed consent form until follow up visit.
* Body mass index (BMI): 18 to 34 kg/m2 (both inclusive);
* Age: 18 to 79 years (both inclusive) at the screening visit;
* Men must agree to use adequate contraception when being sexually active. This applies from signing of the informed consent until 12 weeks after the last study drug administration. 'Adequate contraception' is defined as any combination of at least 2 effective methods of birth control, of which at least one is a physical barrier (e.g. condoms with hormonal contraception or implants or combined oral contraceptives, certain intrauterine devices);
* Ability to understand and follow study-related instructions.

Participants with hepatic impairment

* Participants with documented liver cirrhosis confirmed by histopathology, e.g., previous liver biopsy, laparoscopy, ultrasound, or fibroscan;
* Participants with hepatic impairment (Child Pugh A or B);
* Participants with stable liver disease in the last 2 months.

Healthy participants

* Healthy male and female white participants;
* Mean age and body weight in the control group and in the two groups with hepatic impairment (Child Pugh A and B) should not vary by more than +/-10 years and +/-10 kg;
* Gender matched.

Exclusion Criteria:

All participants

* Participants with a medical disorder, condition, or history of such that would impair the participant's ability to participate or complete this study in the opinion of the investigator or the sponsor;
* Medical history of Kock pouch (ileostomy after proctocolectomy);
* Febrile illness within 1 week prior to admission to study center;
* Relevant diseases within the last 4 weeks prior to admission;
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies;
* Known hypersensitivity to the study drugs;
* Participants with diagnosed malignancy within the past 5 years;
* Participants with psychiatric disorders which may disable the participants to consent;
* Use of the following co-medications from 2 weeks before until 4 days after study drug administration:

  * CYP3A4 inducers (e.g. St. John´s wort, rifampicin, carbamazepin, phenytoin, phenobarbital, bosentan, efavirenz, etravirine, nevirapine)
  * weak to moderate CYP3A4 inhibitors (e.g. grapefruit juice and other grapefruit containing products, erythromycin, saquinavir, amiodarone, verapamil, fluconazole, diltiazem)
  * strong inhibitors of CYP3A4 (e.g. itraconazole, ketoconazol, posaconazole, voriconazole, atazanavir, ritonavir, nelfinavir or other inhibitors of human immunodeficiency virus (HIV) protease, clarithromycin, telithromycin, nefazodon, telaprevir, boceprevir) or
  * gemfibrozil (a strong inhibitor of CYP2C8)
* Positive urine drug screening;
* For women of childbearing potential: positive pregnancy test;
* Positive results for human immunodeficiency virus 1 and 2 antibodies (HIV-Ag/Ab).

Participants with hepatic impairment

* Severe cerebrovascular or cardiac disorders, e.g., myocardial infarction less than 6 months prior to dosing, congestive heart failure of New York Heart Association grade III or IV, severe arrhythmia requiring antiarrhythmic treatment;
* Evidence of hepatic encephalopathy related to chronic liver disease >grade 2 (exclusion by Number Connection Test (NCT);
* Participants with percutaneous transluminal coronary angioplasty or coronary artery bypass graft less than 6 months prior to study drug administration;
* History of bleeding within the past 3 months;
* Thrombotic disorder;
* Participants with diabetes mellitus with a glycohemoglobin A1c (HbA1c) >10%;
* Severe ascites of more than 6 L (estimated by ultrasound);
* Participants with primary and secondary biliary cirrhosis;
* Participants with sclerosing cholangitis;
* Failure of any other major organ system other than the liver;
* Severe infection, malignancy, or psychosis, or any clinically significant illness within 4 weeks prior to study drug administration.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2014-09-16 (Actual); Study Completion 2014-12-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve from zero to infinity (AUC) of finerenone in plasma | 0 hour pre-dose to 96 hour post-dose
Area under the concentration versus time curve from zero to infinity of unbound finerenone (AUCu) in plasma | 0 hour pre-dose to 96 hour post-dose
Maximum observed drug concentration (Cmax) of finerenone in plasma | 0 hour pre-dose to 96 hour post-dose
Maximum observed drug concentration of unbound finerenone (Cmax,u) in plasma | 0 hour pre-dose to 96 hour post-dose

SECONDARY OUTCOMES:
Number of participants with adverse events | From the start of study treatment up to 3 days after study treatment

OTHER OUTCOMES:
Percentage of fraction of free (unbound) (fu) finerenone in plasma | 1 hour post-dose
Area under the concentration versus time curve from zero to infinity divided by dose per kilogram body weight (AUCnorm) of finerenone in plasma | 0 hour pre-dose to 96 hour post-dose
Maximum observed drug concentration divided by dose per kilogram body weight (Cmax,norm) of finerenone in plasma | 0 hour pre-dose to 96 hour post-dose
Time to reach maximum concentration (tmax) of finerenone | 0 hour pre-dose to 96 hour post-dose
Half-life associated with the terminal slope (t1/2) of finerenone | 0 hour pre-dose to 96 hour post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Result] Heinig R, Lambelet M, Nagelschmitz J, Alatrach A, Halabi A. Pharmacokinetics of the Novel Nonsteroidal Mineralocorticoid Receptor Antagonist Finerenone (BAY 94-8862) in Individuals with Mild or Moderate Hepatic Impairment. Eur J Drug Metab Pharmacokinet. 2019 Oct;44(5):619-628. doi: 10.1007/s13318-019-00547-x. PMID 30825073